CLINICAL TRIAL: NCT03857906
Title: Evaluation of Prophylactic Use of a Preoperative Intra-Aortic Ballon Pump in High-Risk Coronary Artery Bypass Graft Surgery: A Single-Centre Study
Brief Title: Evaluation of Prophylactic Use of a Preoperative IABP in High-Risk Coronary Artery Bypass Graft Surgery
Acronym: IABP-HR
Status: Completed | Type: Observational
Sponsor: CMN "20 de Noviembre" (Other)
Collaborators: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Héctor Hugo Escutia Cuevas, Clinical Professor, CMN "20 de Noviembre"
Other Study IDs: .2018
Record Dates: First submitted 2019-02-23; First posted 2019-02-28 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Cardiomyopathy; Heart Failure
Keywords: intra-aortic balloon pump; coronary artery bypass graft; preoperative
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- IABP group: Over 18 years With ischemic heart disease Multivessel disease with/without LMCA involvement High-risk coronary disease Intra-Aortic Ballon Pump insertion 1-6 hours prior to surgery
  Interventions: Device: Intra-Aortic Ballon Pump insertion
- No-IABP group: Over 18 years With ischemic heart disease Multivessel disease with/without LMCA involvement High-risk coronary disease No IABP

INTERVENTIONS:
Device: Intra-Aortic Ballon Pump insertion — The IABP (Ultraflex IAB 7.5F, 2.5mm; Arrow International, Reading, PA) was inserted percutaneously through the right femoral artery in the previous 1 - 6 hours before the scheduled surgery. Positioning of the IABP was guided by radioscopy. The balloon size was based on the patient's height (30, 40 or 50 cc). Transesophageal echocardiography was used to confirm correct IABP placement before and after CABG
  Groups: IABP group

SUMMARY:
Background: The intra-aortic balloon balloon pump (IABP) has been used as a method of percutaneous circulatory assistance high surgical risk patients undergoing coronary artery bypass graft surgery (CABG); Although its applicability has been questioned by clinical trials showing poor impact to reduce the mortality due to cardiogenic shock associated with postoperative acute myocardial infarction (AMI), the real benefit reducing mortality in the postoperative context (PO) has not been determined examined through a prospective study with an adequate design.

Objective: To compare PO complications such as mortality, perioperative infarction and other complications in patients with high surgical risk undergoing CABG in comparison with controls.

DETAILED DESCRIPTION:
Methods: Quasi-experimental, prospective, comparative, non-randomized study. The decision to place the BIAC is not part of the study and depends on the multidisciplinary decision of a Heart Team, based on the individualized risk / benefit. The study population consists on high surgical risk patients with atherosclerotic coronary disease undergoing CABG in our centre between 2014-2018. Patients are excluded if any condition is present: cardiogenic shock, with AMI 48 hours prior and / or severe aortic insufficiency. In one group BIAC will be inserted 1-6 hours before surgery (BIAC group) and a second group is control (non-BIAC group). A minimum 30-day postoperative follow-up of will be performed, with primary end points (mortality and AMI type V) and secondary end points (additional PO complications).

Analysis: An evaluation of normality distribution K-S will be performed, the means of quantitative (t-Test) and categorical variables (Fisher or χ² Pearson) will be compared. A multivariate analysis will be performed with linear logistic regression to evaluate the influence of age, sex, peripheral arterial disease (PAD) and EuroSCORE-II on the primary goal. Statistical significance will be considered when p <0.05. Softwares: GraphPad-Prism-5.0 and SPSS-15.0

ELIGIBILITY:
Inclusion Criteria:

* All patients greater than 18 years
* Scheduled for coronary artery bypass graft (CABG) surgery were eligible
* Multiple vessel disease with or without left main coronary artery (LMCA) significant stenosis (>50%)
* Written informed consent provided

Exclusion Criteria:

* Prior cardiogenic shock,
* Acute myocardial infarction (AMI) less than 48 hours prior to enrollment
* Previous IABP use
* AMI mechanical complications
* Aortic regurgitation greater than grade II in severity (on a scale of I to IV, with higher grades indicating more severe regurgitation)
* Tachyarrhythmia
* Other aortic procedures
* Other non-CABG surgical procedures
* Massive pulmonary embolism
* Older than 90 years of age
* Any coagulopathy
* Severe concomitant disease associated with a life expectancy of less than 6 months.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery were assessed for the inclusion/exclusion criteria, provided signed informed consent, and were allocated to one of two treatments: IABP insertion before skin incision (IABP group) or no IABP insertion (control group). In all cases, the decision of the IABP insertion was generated in a previous Heart Team session, this team was integrated by a Clinical Cardiologist, Cardiac Interventionist, Cardiothoracic Surgeon and Anesthesiologist, in base on the personal risk/benefit of each patient. There was no blinding for patients or physicians in aware of the Heart Team decisions. Outcome assessors were unaware of the assigned treatment.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
30-Day All-Cause Mortality | 30 days
  30-Day Mortality
30-Day Postoperative Myocardial Infarction | 30 days
  Based on the third universal definition on MI criteria

SECONDARY OUTCOMES:
30-day occurrence rate of PCI | 30 days
  30-day occurrence rate of emergent percutaneous coronary intervention
Requirement of mechanical ventilation | 30 days
  Requirement of mechanical ventilation for longer than 24 hours
acute kidney injury | 30 days
  AKIN classification
Need for renal replacement therapy | 30 days
  Need for RRT (hemodialysis, peritoneal)
ICU length of stay | 30 days
  ICU and in-hospital length of stay
Postoperative use of inotropes and vasopressors | 30 days
  Postoperative use of inotropes and vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Juán Antonio Suárez-Cuenca, Principal Investigator — CMN "20 de Noviembre"